CLINICAL TRIAL: NCT03990922
Title: Continuous Thoracic Paravertebral Block for Open Hepatectomy
Brief Title: CTPVB for Hepatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cui Xulei (Other)
Responsible Party: Sponsor-Investigator, Cui Xulei, attending physician, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PVB_H
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Pain Management; Paravertebral Block; Hepatectomy
MeSH Terms: conditions — Agnosia | interventions — Ropivacaine; Sodium Chloride; Analgesia, Patient-Controlled; Morphine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTPVB with ropivocaine (Experimental): Continuous Paravertebral block with ropivacaine and Patient-controlled analgesia with morphine
  Interventions: Procedure: Continuous Paravertebral block with ropivacaine; Drug: Patient-controlled analgesia with morphine
- CTPVB with saline (Placebo Comparator): Continuous Paravertebral block with saline and Patient-controlled analgesia with morphine
  Interventions: Procedure: Continuous Paravertebral "block" with saline; Drug: Patient-controlled analgesia with morphine

INTERVENTIONS:
Procedure: Continuous Paravertebral block with ropivacaine — Inject 25 ml 0.5% ropivacaine in the T8 paravertebral space followed with catheter insertion and continuous 0.2% ropivacaine infusion(infusion rate: 0.125ml/kg/pulse,1pulse/h).
  Arms: CTPVB with ropivocaine
Procedure: Continuous Paravertebral "block" with saline — Inject 25 ml 0.9% saline in the T8 paravertebral space followed with catheter insertion and continuous 0.9% ropivacaine infusion(infusion rate: 0.125ml/kg/pulse,1pulse/h).
  Arms: CTPVB with saline
Drug: Patient-controlled analgesia with morphine — Morphine given as intravenous patient-controlled analgesia bolus: 2mg, lock time: 5min, 1h limitation: 8mg

SUMMARY:
Moderate to severe postoperative pain often influence patients quality of recovery after hepatectomy. Systemic opioids given with patient-controlled analgesia has been used after hepatectomy in many medical center, but the analgesic effect can be limited and undesirable side effects may bring about negative effects on patients recovery. Regional block has been proved to improve patients postoperative recovery in many kinds of surgeries.

The investigators therefore designed a prospective, randomized, subject and assessor blinded, parallel-group, placebo controlled study to test the hypothesis that continuous right thoracic paravertebral block increase patients quality of recovery score on the 7th postoperative day after hepatectomy in patients receiving i.v. patient-controlled analgesia (PCA) with morphine.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 yrs
* American Society of Anesthesiologists physical statusⅠ-Ⅲ
* Undergo hepatectomy with J-shape subcostal incision
* Informed consent

Exclusion Criteria:

* A known allergy to the drugs being used
* Coagulopathy, on anticoagulants
* Analgesics intake, history of substance abuse
* Participating in the investigation of another experimental agent
* Inability to properly describe postoperative pain to investigators (eg, language barrier, neuropsychiatric disorder)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2019-11-09 (Actual); Study Completion 2019-11-17 (Actual)

PRIMARY OUTCOMES:
the postoperative recovery quality on postoperative day 7 | at the 7th postoperative day
  The postoperative recovery quality is evaluated with QoR-15 questionnaire. The QoR-15 is a 15-item questionnaire intended to measure QoR after anesthesia and surgery. It comprises five subscales: pain (2 items), physical comfort (5 items), physical independence (2 items), psychological support (2 items), and emotional state (4 items) [2 Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR- 15. Anesthesiology. 2013;118(6):1332.]. Each item is scored from 0 to 10, and the possible total score ranges from 0(extremely poor quality of recovery) to 150 (excellent quality of re covery).

SECONDARY OUTCOMES:
the postoperative recovery quality on postoperative day 3 | at the 3th postoperative day
  QoR-15 questionnaire The postoperative recovery quality is evaluated with QoR-15 questionnaire. The QoR-15 is a 15-item questionnaire intended to measure QoR after anesthesia and surgery. It comprises five subscales: pain (2 items), physical comfort (5 items), physical independence (2 items), psychological support (2 items), and emotional state (4 items) [2 Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR- 15. Anesthesiology. 2013;118(6):1332.]. Each item is scored from 0 to 10, and the possible total score ranges from 0(extremely poor quality of recovery) to 150 (excellent quality of re covery).
The pain scores determined by the numeric rating scale (NRS, 0-10) | At 8, 24,48 hours after the surgery
  The patients evaluated their pain severity with thenumeric rating scale (NRS, 0-10),where 0 indicates no pain, and 10 indicates the most severe pain
cumulated morphine consumption | At 8, 24,48 hours after the surgery
time to resumption of bowel movement | Up to 2 weeks after surgery
time to out-of bed activity/ambutation | Up to 2 weeks
post operative length of stay | Up to 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: xulei cui, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China